CLINICAL TRIAL: NCT02875366
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design Study of the Effect of Lumacaftor/Ivacaftor Combination Therapy on Exercise Tolerance in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: A Study of the Effects of Lumacaftor/Ivacaftor (LUM/IVA) on Exercise Tolerance in Subjects With Cystic Fibrosis (CF), Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: VX15-809-112; 2016-000066-34 (EudraCT Number)
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to LUM/IVA fixed-dose combination tablet orally every 12 hours (q12h) for 24 weeks.
  Interventions: Drug: Placebo
- LUM/IVA (Experimental): LUM 400 milligram (mg)/IVA 250 mg fixed-dose combination tablet orally q12h for 24 weeks.
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA
  Other Names: Lumacaftor/Ivacaftor
  Arms: LUM/IVA
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 4, randomized, double-blind, placebo-controlled, parallel-group study in subjects aged 12 years and older with CF who are homozygous for the F508del-CFTR mutation. This study is designed to evaluate the effect of LUM/IVA on exercise tolerance in subjects with CF, homozygous for the F508del-CFTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for the F508del-CFTR mutation
* Confirmed diagnosis of CF defined as a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis
* Stable CF disease as judged by the investigator
* Forced expiratory volume in 1 second (FEV1) at least 40% and not greater than 90% of predicted

Exclusion Criteria:

* History of any comorbidity that might confound the results of the study, interfere with the use of cardiopulmonary exercise tests (CPETs) as an assessment, or pose an additional risk in administering study drug to the subject
* Any previous exposure to LUM or IVA
* History of cardiac arrhythmia, ischemic heart disease, congestive heart failure, or other clinically significant cardiac condition, or medical condition requiring chronic use of a beta blocker, non-dihydropyridine calcium channel blocker, or other cardiac medication known to affect exercise tolerance
* History of solid organ or hematological transplantation
* For subjects under 18 years of age at Screening, except those who have had bilateral lens removal, selected findings on a screening ophthalmologic examination will be exclusionary
* Using or expected to require any concomitant medication that is prohibited in this study
* History of alcohol or drug abuse, as deemed by the investigator, in the past year, including but not limited to cannabis, cocaine, and opiates
* Participation in an investigational drug study within 30 days before the Screening Visit
* Pregnant or nursing females; males with a female partner who is pregnant or nursing
* Colonization with organisms associated with a more rapid decline in pulmonary status

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (11):
  - Melbourne, Victoria
  - Parkville, Victoria
  - Adelaide
  - Camperdown
  - Clayton
  - Nedlands
  - New Lambton Heights
  - Randwick
  - South Brisbane
  - Subiaco
  - Westmead
- Edinburgh, United Kingdom

REFERENCES:
- [Derived] Wilson J, You X, Ellis M, Urquhart DS, Jha L, Duncan M, Tian S, Harris RA, Kotsimbos T, Keating D. VO2max as an exercise tolerance endpoint in people with cystic fibrosis: Lessons from a lumacaftor/ivacaftor trial. J Cyst Fibros. 2021 May;20(3):499-505. doi: 10.1016/j.jcf.2020.12.006. Epub 2020 Dec 24. PMID 33358691

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to lumacaftor (LUM)/ivacaftor (IVA) fixed-dose combination tablet orally every 12 hours (q12h) for 24 weeks.
- LUM/IVA: Participants received LUM 400 milligram (mg)/IVA 250 mg fixed-dose combination tablet orally q12h for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | LUM/IVA
Started | 36 | 34
Completed | 36 | 31
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo matched to LUM/IVA fixed-dose combination tablet orally q12h for 24 weeks.
- LUM/IVA: Participants received LUM 400 mg/IVA 250 mg fixed-dose combination tablet orally q12h for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | LUM/IVA | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (10.58) | 24.9 (10.17) | 25.5 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 18 | 21 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 34 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative (Percent) Change From Baseline in Maximal Oxygen Consumption (VO2max) During Cardiopulmonary Exercise Testing (CPET) at Week 24
Description: CPET was used to assess change in exercise tolerance, as measured by VO2max.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) included all randomized participants who received any amount of study drug. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
percent change | -3.5 [-7.7 to 0.8] | -6.6 [-11.3 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.3021, Mixed effects model for repeated measure; Least Squares Mean Difference = -3.2, 95% CI 2-sided [-9.2 to 2.9]

2. Secondary Outcome: Relative (Percent) Change From Baseline in Exercise Duration During CPET at Week 24
Description: Exercise duration is defined as the time at the termination of CPET exercise minus the corresponding time when CPET starts for each CPET exercise.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
percent change | 0.4 [-3.0 to 3.8] | -2.8 [-6.5 to 1.0]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.1894, Mixed effects model for repeated measure; Least Squares Mean Difference = -3.2, 95% CI 2-sided [-8.0 to 1.6]

3. Secondary Outcome: Absolute Change From Baseline in Exercise Duration During CPET at Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
seconds | -2.1 [-20.0 to 15.9] | -17.4 [-37.2 to 2.4]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.2328, Mixed effects model for repeated measure; Least Squares Mean Difference = -15.3, 95% CI 2-sided [-40.8 to 10.1]

4. Secondary Outcome: Absolute Change From Baseline in VO2max During CPET at Week 24
Description: CPET was used to assess change in exercise tolerance, as measured by VO2max.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per kilogram per minute
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
milliliter per kilogram per minute | -1.3 [-2.5 to -0.1] | -2.7 [-4.0 to -1.3]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.1203, Mixed effects model for repeated measure; Least Squares Mean Difference = -1.4, 95% CI 2-sided [-3.1 to 0.4]

5. Secondary Outcome: Absolute Change From Baseline in Oxygen Consumption (VO2) at Anaerobic Threshold at Week 24
Description: Anaerobic threshold was defined as the exercise intensity at which lactate starts to accumulate.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per minute
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 25
milliliter per minute | 94.6 [-5.8 to 195.0] | -55.1 [-168.0 to 57.9]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.0439, Mixed effects model for repeated measure; Least Squares Mean Difference = -149.6, 95% CI 2-sided [-295.0 to -4.2]

6. Secondary Outcome: Relative (Percent) Change From Baseline in VO2 at Anaerobic Threshold at Week 24
Description: Anaerobic threshold was defined as the exercise intensity at which lactate starts to accumulate.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 25
percent change | 9.4 [0.9 to 17.8] | 1.8 [-7.7 to 11.3]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.2237, Mixed effects model for repeated measure; Least Squares Mean Difference = -7.5, 95% CI 2-sided [-19.8 to 4.7]

7. Secondary Outcome: Absolute Change From Baseline in Functional VO2 Gain at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliter per minute per watt
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
milliliter per minute per watt | 0.07 [-0.29 to 0.43] | -0.53 [-0.93 to -0.14]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.0226, Mixed effects model for repeated measure; Least Squares Mean Difference = -0.60, 95% CI 2-sided [-1.12 to -0.09]

8. Secondary Outcome: Relative (Percent) Change From Baseline in Functional VO2 Gain at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 26
percent change | 1.46 [-3.10 to 6.03] | -4.85 [-9.93 to 0.22]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.0613, Mixed effects model for repeated measure; Least Squares Mean Difference = -6.32, 95% CI 2-sided [-12.94 to 0.31]

9. Secondary Outcome: Absolute Change From Baseline in Pulmonary Ventilation (VE) Versus Carbon Dioxide Production (VCO2) Slope at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 31 | 26
ratio | 0.5 [-0.3 to 1.4] | 0.8 [-0.1 to 1.7]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.6409, Mixed effects model for repeated measure; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-0.9 to 1.5]

10. Secondary Outcome: Relative (Percent) Change From Baseline in Pulmonary Ventilation (VE) Versus Carbon Dioxide Production (VCO2) Slope at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 31 | 26
percent change | 2.0 [-0.7 to 4.6] | 3.0 [0.1 to 5.8]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.5889, Mixed effects model for repeated measure; Least Squares Mean Difference = 1.0, 95% CI 2-sided [-2.7 to 4.7]

11. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted FEV1
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 30
percentage of predicted FEV1 | -4.0 [-7.3 to -0.7] | -0.6 [-4.0 to 2.9]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.1460, Mixed effects model for repeated measure; Least Squares Mean Difference = 3.4, 95% CI 2-sided [-1.2 to 8.1]

12. Secondary Outcome: Relative (Percent) Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 32 | 30
percent change | -5.4 [-10.3 to -0.5] | -1.8 [-6.9 to 3.2]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.3091, Mixed effects model for repeated measure; Least Squares Mean Difference = 3.5, 95% CI 2-sided [-3.4 to 10.4]

13. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 24
Description: BMI was defined as weight in kilograms (kg) divided by height in square meter (m^2).
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 33 | 30
kg/m^2 | 0.3 [0.0 to 0.6] | 0.5 [0.1 to 0.8]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.3961, Mixed effects model for repeated measure; Least Squares Mean Difference = 0.2, 95% CI 2-sided [-0.3 to 0.6]

14. Secondary Outcome: Relative (Percent) Change From Baseline in BMI at Week 24
Description: BMI was defined as weight in kg divided by height in m^2.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 33 | 30
percent change | 1.5 [0.0 to 3.1] | 2.5 [0.9 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.3905, Mixed effects model for repeated measure; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-1.2 to 3.1]

15. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score at Week 24
Description: The CFQ-R assessed respiratory symptoms on a scale with scores ranging from 0 to 100; where higher scores indicated fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 33 | 30
units on a scale | -6.1 [-11.7 to -0.5] | 0.1 [-5.9 to 6.1]
Statistical Analysis 1: Comparison: Placebo vs LUM/IVA; Test type: Superiority; p = 0.1257, Mixed effects model for repeated measure; Least Squares Mean Difference = 6.2, 95% CI 2-sided [-1.8 to 14.1]

16. Secondary Outcome: Number of Participants in Each Severity Category of Patient Health Questionnaire (PHQ-8)
Description: The PHQ-8 is an eight item self-reported measure of depression. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Total score is the sum of individual eight items and ranges from 0 to 24, with higher scores indicating more severe depression symptoms. Total score of 0 to 5 indicates none to minimal depression, 6 to 10 indicates mild depression, 11 to 15 indicates moderate depression, 16 to 20 indicates moderately severe depression and 21 to 24 indicates severe depression.
Time Frame: Baseline, Week 24
Population: FAS. Here "Number Analyzed" signifies those participants who were evaluated for this outcome at the specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 36 | 34
participants
  Baseline: None to minimal | 27 | 28
  Baseline: Mild | 8 | 5
  Baseline: Moderate | 0 | 1
  Baseline: Moderately severe | 1 | 0
  Baseline: Severe | 0 | 0
  Week 24: None to minimal: number analyzed (Participants) | 33 | 30
  Week 24: None to minimal | 23 | 24
  Week 24: Mild: number analyzed (Participants) | 33 | 30
  Week 24: Mild | 8 | 3
  Week 24: Moderate: number analyzed (Participants) | 33 | 30
  Week 24: Moderate | 1 | 3
  Week 24: Moderately severe: number analyzed (Participants) | 33 | 30
  Week 24: Moderately severe | 1 | 0
  Week 24: Severe: number analyzed (Participants) | 33 | 30
  Week 24: Severe | 0 | 0

17. Secondary Outcome: Number of Participants in Each Severity Category of Generalized Anxiety Disorder (GAD-7) Scores
Description: The GAD-7 is a seven item, self-reported measurement of GAD severity. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Total score is the sum of individual seven items and ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms. Total score of 0 to 5 indicates none to minimal anxiety, 6 to 10 indicates mild anxiety, 11 to 15 indicates moderate anxiety, 16 to 21 indicates severe anxiety.
Time Frame: Baseline, Week 24
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 36 | 34
participants
  Baseline: None to minimal | 31 | 29
  Baseline: Mild | 5 | 5
  Baseline: Moderate | 0 | 0
  Baseline: Severe | 0 | 0
  Week 24: None to minimal: number analyzed (Participants) | 33 | 30
  Week 24: None to minimal | 26 | 26
  Week 24: Mild: number analyzed (Participants) | 33 | 30
  Week 24: Mild | 6 | 3
  Week 24: Moderate: number analyzed (Participants) | 33 | 30
  Week 24: Moderate | 1 | 1
  Week 24: Severe: number analyzed (Participants) | 33 | 30
  Week 24: Severe | 0 | 0

18. Secondary Outcome: Absolute Change From Baseline in Daily Physical Activity Counts as Determined by Actigraphy at Week 24
Description: Participants were provided with a wrist-worn actigraphy device which continuously collected data about daily physical activity counts.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: physical activity counts per day
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 19 | 20
physical activity counts per day | -23239 (73936.4) | -22409 (52450.1)

19. Secondary Outcome: Relative (Percent) Change From Baseline in Physical Activity as Determined by Actigraphy at Week 24
Description: Participants were provided with a wrist-worn actigraphy device which continuously collected data about daily physical activities.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 19 | 20
percent change | -5 (26.9) | -7 (24.3)

20. Secondary Outcome: Absolute Change From Baseline in Duration of Sleep Time at Week 24
Description: Participants were provided with a wrist-worn actigraphy device which continuously collected data about sleep duration and quality.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 18 | 18
hours | -0.4 (0.88) | 0.1 (0.74)

21. Secondary Outcome: Relative (Percent) Change From Baseline in Duration of Sleep Time at Week 24
Description: as for outcome 20
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 18 | 18
percent change | -5.7 (12.30) | 1.5 (9.79)

22. Secondary Outcome: Absolute Change From Baseline in Time Above Sedentary Duration at Week 24
Description: Participants were provided with a wrist-worn actigraphy device which continuously collected data about daily activities and sleep duration and quality.
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 15 | 21
hours | -0.7 (1.48) | -0.7 (2.09)

23. Secondary Outcome: Relative (Percent) Change From Baseline in Time Above Sedentary Duration at Week 24
Description: as for outcome 22
Time Frame: Baseline, Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 15 | 21
percent change | 0.2 (64.76) | 2.3 (77.18)

24. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 28
Population: The Safety Set was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LUM/IVA
Number analyzed (Participants) | 36 | 34
participants
  Participants With AEs | 35 | 30
  Participants With SAEs | 9 | 15

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Arm/Group | Placebo | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 9/36 | 15/34
Other Adverse Events (participants affected / at risk) | 34/36 | 28/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | LUM/IVA (N=34)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 6 | 8
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | LUM/IVA (N=34)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 5 | 3
Toothache (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Bacterial test positive (Investigations) | 2 | 0
Blood iron decreased (Investigations) | 2 | 0
Fungal test positive (Investigations) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT02875366/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT02875366/SAP_001.pdf